CLINICAL TRIAL: NCT01669135
Title: Spinal Anesthesia for Cesarean Delivery is Associated With Decreases in Regional Cerebral Oxygen Saturation as Assessed by Near- Infrared Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, MD, PhD, DEAA, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M19-12-21-2010
Record Dates: First submitted 2012-08-08; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Cerebral Oxygen Saturation During Spinal Anesthesia for Cesarean Delivery
Keywords: cerebral oximetry; cesarean delivery
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Anesthesia with cerebral oxygen saturation monitoring (Other): The cerebral oxygen saturation of the right and left frontal lobe as well as the thigh oxygen saturation are monitored during spinal anesthesia by means of the near-infrared spectroscopy. Hemodynamic variables were recorded at the same time points.
  Interventions: Other: Spinal Anesthesia with cerebral oxygen saturation monitoring

INTERVENTIONS:
Other: Spinal Anesthesia with cerebral oxygen saturation monitoring
  Other Names: INVOS (cerebral oximeter model 5100, Somanetics, Troy, MI, USA)

SUMMARY:
The cerebral oxygen saturation is assessed by means of near-infrared spectometry in parturients undergoing cesarean delivery under spinal anesthesia. The investigators hypothesis was that spinal anesthesia does not influence cerebral oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Term healthy parturients

Exclusion Criteria:

* Body Mass Index > 35
* preeclampsia
* neurological,cardiovascular, respiratory disease

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
cerebral oxygen saturation of the right frontal lobe | Change from the performing of spinal anesthesia untill 1 minute after delivery
  Cerebral oxygen saturation is important as it may affect patient's outcome

SECONDARY OUTCOMES:
cerebral oxygen saturation of the left frontal lobe | 5, 10, 50 min after spinal,1 minute after delivery
  Cerebral oxygen saturation is important for patient's outcome
Thigh oxygen saturation | 5, 10, 50 min after spinal, 1 minute after delivery
  Thigh oxygen saturation may reflect blood redistribution due to spinal block
Arterial Oxygenation | 5, 10, 50 min after spinal, 1 minute after delivery
  Changes in arterial oxygenation may reflect blood redistribution due to spinal block

OTHER OUTCOMES:
Hemodynamic changes (Changes in Blood Pressure (mmHg) and Heart rate (beats/min) | 5, 10, 50 min after spinal, 1 minute after delivery
  Hemodynamic changes (changes in Blood Pressure and Heart rate) may reflect blood redistribution due to spinal block

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Aretaieio Hospital, Athens, Greece

REFERENCES:
- [Derived] Fassoulaki A, Paraskeva A, Tsaroucha A. Cesarean delivery under spinal anesthesia is associated with decreases in cerebral oxygen saturation as assessed by NIRS: an observational study. Curr Med Res Opin. 2014 Mar;30(3):331-7. doi: 10.1185/03007995.2013.852526. Epub 2013 Nov 8. PMID 24106922